CLINICAL TRIAL: NCT06311305
Title: Does Early Laparoscopic Cholecystectomy After ERCP Reduce the Risk of Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdulla Mohammed Ahmed, Abdulla Mohammed Ahmed Hussein, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-med-24-03-07MS
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cholelithiases
Keywords: ERCP; Laparoscopic; cholecystectomy; Gallstones
MeSH Terms: conditions — Cholelithiasis; Gallstones | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: we aim to assess if the early laparoscopic cholecystectomy after ERCP can reduce the risks or complications
Masking Description: NONE (open label single group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- early laparoscopic cholecystectomy after ERCP (Other): we assess the risks and complications of early laparoscopic cholecystectomy after ERCP
  Interventions: Procedure: Early Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Early Laparoscopic cholecystectomy — laparoscopic cholecystectomy early after ERCP with assessing the risks and complications
  Other Names: laparoscopic cholecystectomy

SUMMARY:
Gallstones have been recognised since antiquity and have been found during autopsies of Egyptian mummies. Following the first successful open cholecystectomy in 1882, it was Eric Muhe, a German surgeon, who performed the first laparoscopic cholecystectomy (Lapara, the flank; and skopein, to examine) in 1985.

The common mechanism of gallstone formation includes cholesterol hypersecretion, alteration in intestinal bile salt, cholesterol absorption and gall bladder hypokinesia, which leads to bile cholesterol supersaturation and nucleation.

Incidence of CBD stones in cases of cholelithiasis is around 3.4%-15%.2 Choledocholithiasis can either be primary or secondary. Secondary Choledocholithiasis being more common occurs due to stones originating in gallbladder and then migrating through cystic duct to CBD. Primary bile duct stones originate from within bile ducts and are more common in Asian populations. These stones are associated with biliary stasis and bacteria.

DETAILED DESCRIPTION:
Gallstones have been recognised since antiquity and have been found during autopsies of Egyptian mummies. Following the first successful open cholecystectomy in 1882, it was Eric Muhe, a German surgeon, who performed the first laparoscopic cholecystectomy (Lapara, the flank; and skopein, to examine) in 1985. 1 The common mechanism of gallstone formation includes cholesterol hypersecretion, alteration in intestinal bile salt, cholesterol absorption and gall bladder hypokinesia, which leads to bile cholesterol supersaturation and nucleation.2 Incidence of CBD stones in cases of cholelithiasis is around 3.4%-15%.2 Choledocholithiasis can either be primary or secondary. Secondary Choledocholithiasis being more common occurs due to stones originating in gallbladder and then migrating through cystic duct to CBD. Primary bile duct stones originate from within bile ducts and are more common in Asian populations. These stones are associated with biliary stasis and bacteria.3 The diagnosis of choledocholithiasis is initially suggested by symptomatology, laboratory tests, and ultrasound (US) findings. Abdominal ultrasound being the most commonly used initial diagnostic tool for suspected biliary stones has a sensitivity of 25-60% and specificity of 95-100%.4 Ultrasound can reliably detect a dilated extrahepatic bile duct, typically a CBD > 6 mm. However, a large study of patients undergoing cholecystectomy found that nearly half of the patients with choledocholithiasis have a nondilated CBD.5 Moreover, the diameter of the extrahepatic bile duct increases with age and older patients may have a normal duct greater than 6 mm. Largely, due to its poor sensitivity, a negative US does not rule out choledocholithiasis. Contrast enhanced computed tomography has a sensitivity of 71-85% and specificity of 88-95% which can further be improved by addition of a hepatobiliary-excreted intravenous contrast agent.6,7 Since the introduction in 1991, Magnetic resonance cholangiopancreatography (MRCP) has emerged as an accurate, non-invasive diagnostic modality for investigating the biliary and pancreatic ducts with sensitivity of 90-100% and specificity of 92-100%.8,9 An impacted biliary stone will appear as a filling defect with a crescent of bile.10 In 1968, ERCP was introduced as a diagnostic tool in the management of biliary and pancreatic diseases.11 With introduction of Endoscopic sphincterotomy, ERCP has now developed as a therapeutic tool with sensitivity of 90% and specificity of 98%.12 ERCP stone extraction is successful 80% - 90% of time using the techniques of sphincterotomy and balloon catheter or Dormia basket stone retrieval.13 Pancreatitis is the most common complication seen after ERCP. ERCP- induced pancreatitis is defined as new or worsened abdominal pain with serum amylase that is greater than three times the upper limit of normal at 24 hours post procedure and requires at least two days of hospitalisation. Although transient elevation of pancreatic enzymes i.e. serum amylase and serum lipase are evident after ERCP.14 Long term complications include papillary stenosis, cholangitis and recurrent choledocholithiasis.15 The introduction of Laparoscopic cholecystectomy has significantly influenced the treatment of patients with gallstones. Currently it is estimated that over 80% of cholecystectomies are performed using the laparoscopic approach. Advantages of laparoscopic cholecystectomy include earlier bowel function, less postoperative pain, improved cosmesis, shorter length of hospital stay, earlier return to full activity and decreased overall cost. Laparoscopic cholecystectomy (LC) preceded by preoperative ERCP remains the cornerstone and most commonly practiced strategy worldwide for the management of coexisting gallbladder and CBD stones.16 According to the literature, the conversion rate for laparoscopic cholecystectomy (LC) after endoscopic sphincterotomy (ES) for choledocholithiasis reaches 20%, when laparoscopic cholecystectomy is performed 6 to 8 weeks afterward3. Also, many Patients waiting to undergo cholecystectomy after ES for CBD stones, experiences recurrent biliary events requiring repeated endoscopic reintervention, emergency cholecystectomy or both which not only have an obvious influence on a patient's well-being, but also appear to be associated with increased difficulty of surgery and a more complicated postoperative course.17.

Cholecystectomy is often performed after ERCP (endoscopic retrograde cholangiopancreatography) for patients with gallstones in the common bile duct. However, cholecystectomy after ERCP may have some risks and complications, such as:

* Longer operative time and increased bleeding
* Higher conversion rate to open cholecystectomy
* Difficulty in achieving the critical view of safety
* More post-operative drain and longer hospital stay
* Infection, perforation, pancreatitis, or bile leak. 17.18 Post ERCP cholecystectomy assessment of difficulty is important to reduce the complications , conversion rate , choose of surgery team ,schedule surgery and improve outcomes .There are multiple risk factor associated with post ERCP cholecystectomyhave beenpreviously described in the literature such as age , sex , obesity anatomical variation ,previous surgery , impacted stone etc .Intra operatively, it has been observed that surgeons encountered difficulty while LC post ERCP when there were dense adhesions at calot's triangle, fibrotic and contracted gallbladder,acutely inflamed or cholecysto-enteric fistula etc.19 The risk of complications may depend on several factors, such as the timing of cholecystectomy after ERCP, the presence of a stent in the bile duct, the severity of gallstone disease, and the experience of the surgeon¹²⁴. Therefore, it is important to discuss the benefits and risks of cholecystectomy after ERCP .20

ELIGIBILITY:
Inclusion Criteria:

* Patients post ERCP with gall stone.
* Age 15-70
* Gender female and male patient.

Exclusion Criteria:

* Post ERCP pancreatitis
* Septicemia
* Hepatocellular jaundice and End stage liver disease
* Patient who didn't give informed consent.
* Patients who refused laparoscopic cholecystectomy.
* Patients who were not fit for general anesthesia due to various medical illnesses.
* ERCP for reasons other than stone disease,
* Contraindications to Laparoscopic cholecystectomy like: Cardiovascular andpulmonary disease, coagulopathies and end-stage liver disease (ESLD).
* Patients with Carcinoma Gall bladder, Common bile duct strictures, Coagulopathy, previous upper abdominal surgeries

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
bile leakage | 2 weeks postoperative
  yes or no
operative time | intraoperative
  in hours
intraoperative bleeding | intraoperative
  in cubic centimeters
sepsis | 2 weeks postoperative
  yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No